CLINICAL TRIAL: NCT02587520
Title: Safety and Immunogenicity of Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed (SP0173) in Healthy Adolescents, Adults, and Older Adults
Brief Title: Study of Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ADC01; U1111-1161-3027 (Other: WHO)
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Tetanus; Diphtheria; Pertussis; Whooping Cough
Keywords: Tetanus; Diphtheria; Pertussis; SP0173; Tdap vaccine
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (18):
- Adolescents: SP0173 Formulation 1 (Experimental): Healthy participants aged 10-18 years received a single dose of the SP0173 Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed (Tdap) vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed Formulation 1
- Adolescents: SP0173 Formulation 2 (Experimental): Healthy participants aged 10-18 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 2
- Adolescents: SP0173 Formulation 3 (Experimental): Healthy participants aged 10-18 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 3
- Adolescents: SP0173 Formulation 4 (Experimental): Healthy participants aged 10-18 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 4
- Adolescents: Adacel® (Active Comparator): Healthy participants aged 10-18 years received Adacel®.
  Interventions: Biological: Licensed Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed
- Adolescents: Boostrix® (Active Comparator): Healthy participants aged 10-18 years received Boostrix®.
  Interventions: Biological: Licensed Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine
- Adults: SP0173 Formulation 1 (Experimental): Healthy participants aged 19-64 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed Formulation 1
- Adults: SP0173 Formulation 2 (Experimental): Healthy participants aged 19-64 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 2
- Adults: SP0173 Formulation 3 (Experimental): Healthy participants aged 19-64 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 3
- Adults: SP0173 Formulation 4 (Experimental): Healthy participants aged 19-64 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 4
- Adults: Adacel® (Active Comparator): Healthy participants aged 19-64 years received Adacel®.
  Interventions: Biological: Licensed Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed
- Adults: Boostrix® (Active Comparator): Healthy participants aged 19-64 years received Boostrix®.
  Interventions: Biological: Licensed Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine
- Older Adults: SP0173 Formulation 1 (Experimental): Healthy participants aged greater than equal to (>=65) years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed Formulation 1
- Older Adults: SP0173 Formulation 2 (Experimental): Healthy participants aged >=65 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 2
- Older Adults: SP0173 Formulation 3 (Experimental): Healthy participants aged >=65 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 3
- Older Adults: SP0173 Formulation 4 (Experimental): Healthy participants aged >= 65 years received a single dose of the SP0173 Tdap vaccine.
  Interventions: Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 4
- Older Adults: Adacel® (Active Comparator): Healthy participants aged >=65 years received Adacel®.
  Interventions: Biological: Licensed Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed
- Older Adults: Boostrix® (Active Comparator): Healthy participants aged >=65 years received Boostrix®.
  Interventions: Biological: Licensed Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine

INTERVENTIONS:
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed Formulation 1 — 0.5 milliliter (mL), Intramuscular
  Other Names: SP0173
  Arms: Adolescents: SP0173 Formulation 1; Adults: SP0173 Formulation 1; Older Adults: SP0173 Formulation 1
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 2 — 0.5 mL, Intramuscular
  Other Names: SP0173
  Arms: Adolescents: SP0173 Formulation 2; Adults: SP0173 Formulation 2; Older Adults: SP0173 Formulation 2
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 3 — 0.5 mL, Intramuscular
  Other Names: SP0173
  Arms: Adolescents: SP0173 Formulation 3; Adults: SP0173 Formulation 3; Older Adults: SP0173 Formulation 3
Biological: Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed, Formulation 4 — 0.5 mL, Intramuscular
  Other Names: SP0173
  Arms: Adolescents: SP0173 Formulation 4; Adults: SP0173 Formulation 4; Older Adults: SP0173 Formulation 4
Biological: Licensed Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine Adsorbed — 0.5 mL, Intramuscular
  Arms: Adolescents: Adacel®; Adults: Adacel®; Older Adults: Adacel®
Biological: Licensed Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine — 0.5 mL, Intramuscular
  Arms: Adolescents: Boostrix®; Adults: Boostrix®; Older Adults: Boostrix®

SUMMARY:
This was a dose and formulation ranging study to assess the safety and immunogenicity of SP0173 in healthy adolescents, adults, and older adults in the United States (US).

Primary Objective

* To describe the safety profile of each SP0173 investigational formulation.

Observational Objective:

* To describe the immunogenicity of each SP0173 investigational formulation.

DETAILED DESCRIPTION:
All participants received a single dose of vaccine, and were assessed for immunogenicity at baseline (pre-vaccination) and at 30 days post-vaccination. They were also monitored for safety from day of vaccination up to Day 180 post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 18 years, 19 to 64 years, or >= 65 years on the day of inclusion.
* Informed consent form had been signed and dated by the participant, or assent form had been signed and dated by the participant and informed consent form had been signed and dated by the parent/guardian
* Participant or participant and parent/guardian able to attend all scheduled visits and to comply with all study procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential, (to be considered of non-childbearing potential, a female must be premenarche or post-menopausal for at least 1 year) surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination.
* Participation at the time of study enrollment or planned participation during the present study period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Received any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine between Visit 1 and Visit 2.
* Known or suspected receipt of a tetanus toxoid, reduced diphtheria toxoid, and Acellular pertussis (Tdap) vaccine or Tdap-containing vaccine at any point in time, or receipt of a tetanus and diphtheria containing vaccine in the preceding 5 years.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* History of diphtheria, tetanus, or pertussis infection (confirmed either serologically or microbiologically).
* Known or suspected systemic hypersensitivity to any of the vaccine components or history of life-threatening reaction to the study vaccine or a vaccine containing the same substances.
* Laboratory-confirmed / self-reported thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* History of encephalopathy (e.g., coma, decreased level of consciousness, or prolonged seizures) not attributable to another identifiable cause within 7 days of administration of a previous dose of diphtheria and tetanus toxoids and pertussis (DTP), or diphtheria and tetanus toxoids and acellular pertussis (DTaP) vaccine.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection on the day of vaccination or febrile illness (temperature >= 100.4°F).
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1363 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (19):
- United States (19):
  - Birmingham, Alabama
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - San Diego, California
  - DeLand, Florida
  - Miami, Florida
  - Orlando, Florida
  - Meridian, Idaho
  - Bardstown, Kentucky
  - Nicholasville, Kentucky
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Rochester, New York
  - Cleveland, Ohio
  - Erie, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 20 centers in the Unites States (US) from 22 October 2015 to 15 August 2016.
Pre-assignment Details: A total of 1363 participants were randomized in a 1:1:1 ratio to 1 of the 6 formulation study groups. Randomization was stratified by age (adolescents: age 10-18 years, adults: age 19-64 years, and older adults: age greater than equal to [>=] 65 years).
Groups:
- Older Adults: SP0173 Formulation 1; Older Adults: SP0173 Formulation 2: Healthy participants aged >=65 years received a single dose of the SP0173 Tdap vaccine.
- Older Adults: SP0173 Formulation 3: Healthy subjects aged >=65 years received a single dose of the SP0173 Tdap vaccine.
- Older Adults: SP0173 Formulation 4: Healthy subjects aged >= 65 years received a single dose of the SP0173 Tdap vaccine.
Period: Overall Study
Arm/Group | Adolescents: SP0173 Formulation 1 | Adolescents: SP0173 Formulation 2 | Adolescents: SP0173 Formulation 3 | Adolescents: SP0173 Formulation 4 | Adolescents: Adacel® | Adolescents: Boostrix® | Adults: SP0173 Formulation 1 | Adults: SP0173 Formulation 2 | Adults: SP0173 Formulation 3 | Adults: SP0173 Formulation 4 | Adults: Adacel® | Adults: Boostrix® | Older Adults: SP0173 Formulation 1 | Older Adults: SP0173 Formulation 2 | Older Adults: SP0173 Formulation 3 | Older Adults: SP0173 Formulation 4 | Older Adults: Adacel® | Older Adults: Boostrix®
Started | 80 | 71 | 78 | 79 | 75 | 75 | 76 | 73 | 76 | 76 | 76 | 73 | 77 | 74 | 78 | 72 | 76 | 78
Safety Analysis Set (SafAS) (All participants who received study vaccine, analyzed according to vaccine actually received.) | 79 | 71 | 77 | 77 | 75 | 75 | 76 | 73 | 76 | 76 | 76 | 72 | 77 | 73 | 78 | 72 | 76 | 78
Completed | 78 | 69 | 77 | 74 | 75 | 72 | 73 | 71 | 73 | 71 | 73 | 69 | 77 | 73 | 78 | 72 | 76 | 78
Not Completed | 2 | 2 | 1 | 5 | 0 | 3 | 3 | 2 | 3 | 5 | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adolescents: SP0173 Formulation 1 | Adolescents: SP0173 Formulation 2 | Adolescents: SP0173 Formulation 3 | Adolescents: SP0173 Formulation 4 | Adolescents: Adacel® | Adolescents: Boostrix® | Adults: SP0173 Formulation 1 | Adults: SP0173 Formulation 2 | Adults: SP0173 Formulation 3 | Adults: SP0173 Formulation 4 | Adults: Adacel® | Adults: Boostrix® | Older Adults: SP0173 Formulation 1 | Older Adults: SP0173 Formulation 2 | Older Adults: SP0173 Formulation 3 | Older Adults: SP0173 Formulation 4 | Older Adults: Adacel® | Older Adults: Boostrix® | Total
Number analyzed (Participants) | 80 | 71 | 78 | 79 | 75 | 75 | 76 | 73 | 76 | 76 | 76 | 73 | 77 | 74 | 78 | 72 | 76 | 78 | 1363
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (1.3) | 11.0 (1.3) | 11.1 (1.6) | 10.8 (1.4) | 10.8 (1.5) | 11.1 (1.6) | 42.5 (12.5) | 41.2 (12.1) | 40.1 (12.8) | 42.1 (13.0) | 41.3 (12.7) | 42.5 (13.2) | 71.3 (5.4) | 71.8 (5.4) | 70.9 (4.8) | 70.8 (5.1) | 70.9 (5.0) | 71.3 (4.8) | 41.2 (25.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 33 | 35 | 37 | 39 | 40 | 43 | 46 | 38 | 39 | 44 | 36 | 37 | 38 | 51 | 38 | 46 | 45 | 726
  Male | 39 | 38 | 43 | 42 | 36 | 35 | 33 | 27 | 38 | 37 | 32 | 37 | 40 | 36 | 27 | 34 | 30 | 33 | 637
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 3 | 4 | 4 | 6 | 17 | 19 | 8 | 11 | 15 | 10 | 11 | 12 | 13 | 15 | 12 | 13 | 179
  Not Hispanic or Latino | 76 | 69 | 75 | 75 | 71 | 69 | 59 | 54 | 68 | 65 | 61 | 63 | 64 | 59 | 64 | 55 | 63 | 61 | 1171
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 2 | 1 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 8
  Asian | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 7 | 9 | 2 | 4 | 8 | 4 | 23 | 18 | 24 | 18 | 23 | 19 | 7 | 8 | 8 | 5 | 6 | 10 | 203
  White | 71 | 60 | 71 | 72 | 63 | 65 | 48 | 51 | 46 | 53 | 52 | 51 | 69 | 64 | 70 | 66 | 69 | 68 | 1109
  More than one race | 2 | 1 | 3 | 2 | 2 | 4 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Injections Site or Systemic Reactions Following Vaccination at Day 0: Aged 10-18 Years
Description: A solicited reaction (SR) is an adverse event (AE) that is prelisted in the electronic Case Report Form (eCRF) and considered to be related to vaccination. An SR is therefore an adverse drug reaction (ADR) observed and reported under the conditions (nature & onset) prelisted (i.e., solicited) in the eCRF. An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or onset post-vaccination. Solicited injection site reactions: Pain, Erythema, Swelling, Upper limb edema, Extensive limb swelling and solicited systemic reactions: Fever, Headache, Malaise, Myalgia. Number of participants with at least one solicited injection site reactions and systemic reactions were reported.
Time Frame: Within 7 days after vaccination
Population: Safety analysis set that was defined as those participants who had received study vaccine. All participants had their safety analyzed according to the vaccine they actually received. Here, "number analyzed"= number of participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents: SP0173 Formulation 1 | Adolescents: SP0173 Formulation 2 | Adolescents: SP0173 Formulation 3 | Adolescents: SP0173 Formulation 4 | Adolescents: Adacel® | Adolescents: Boostrix®
Number analyzed (Participants) | 79 | 71 | 77 | 77 | 75 | 75
Participants
  Injection site pain: number analyzed (Participants) | 78 | 69 | 77 | 74 | 75 | 73
  Injection site pain | 59 | 51 | 50 | 49 | 59 | 48
  Injection site erythema: number analyzed (Participants) | 78 | 69 | 77 | 74 | 75 | 73
  Injection site erythema | 9 | 4 | 10 | 1 | 4 | 2
  Injection site swelling: number analyzed (Participants) | 78 | 69 | 77 | 74 | 75 | 73
  Injection site swelling | 7 | 4 | 8 | 0 | 1 | 4
  Upper limb edema: number analyzed (Participants) | 77 | 69 | 77 | 74 | 74 | 73
  Upper limb edema | 45 | 41 | 49 | 46 | 48 | 33
  Extensive limb swelling | 0 | 0 | 0 | 0 | 0 | 0
  Fever: number analyzed (Participants) | 77 | 69 | 77 | 74 | 75 | 73
  Fever | 1 | 0 | 1 | 0 | 0 | 1
  Headache: number analyzed (Participants) | 78 | 69 | 77 | 74 | 75 | 73
  Headache | 21 | 14 | 19 | 25 | 20 | 27
  Malaise: number analyzed (Participants) | 78 | 69 | 77 | 74 | 75 | 73
  Malaise | 14 | 17 | 14 | 18 | 12 | 17
  Myalgia: number analyzed (Participants) | 78 | 69 | 77 | 74 | 75 | 73
  Myalgia | 42 | 35 | 38 | 42 | 52 | 38

2. Primary Outcome: Number of Participants With Solicited Injections Site or Systemic Reactions Following Vaccination at Day 0: Aged 19-64 Years
Description: An SR is an AE that is prelisted in the eCRF and considered to be related to vaccination. An SR is therefore an ADR observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the eCRF. An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or onset post-vaccination. Solicited injection site reactions: Pain, Erythema, Swelling, Upper limb edema, Extensive limb swelling and systemic reactions: Fever, Headache, Malaise, Myalgia. Number of participants with at least one solicited injection site reactions and systemic reactions were reported.
Time Frame: Within 7 days after vaccination
Population: Analysis was performed on safety analysis set. Here, "number analyzed"=number of participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Adults: SP0173 Formulation 1 | Adults: SP0173 Formulation 2 | Adults: SP0173 Formulation 3 | Adults: SP0173 Formulation 4 | Adults: Adacel® | Adults: Boostrix®
Number analyzed (Participants) | 76 | 73 | 76 | 76 | 76 | 72
Participants
  Injection site pain: number analyzed (Participants) | 73 | 70 | 73 | 71 | 72 | 68
  Injection site pain | 38 | 34 | 49 | 42 | 49 | 35
  Injection site erythema: number analyzed (Participants) | 73 | 70 | 73 | 71 | 72 | 68
  Injection site erythema | 2 | 1 | 2 | 0 | 5 | 2
  Injection site swelling: number analyzed (Participants) | 73 | 70 | 73 | 71 | 72 | 68
  Injection site swelling | 1 | 3 | 4 | 1 | 3 | 1
  Upper limb edema: number analyzed (Participants) | 71 | 67 | 72 | 69 | 71 | 67
  Upper limb edema | 28 | 37 | 41 | 37 | 35 | 31
  Extensive limb swelling | 0 | 0 | 0 | 0 | 1 | 0
  Fever: number analyzed (Participants) | 71 | 68 | 72 | 70 | 71 | 68
  Fever | 0 | 0 | 0 | 0 | 2 | 1
  Headache: number analyzed (Participants) | 73 | 71 | 73 | 71 | 72 | 68
  Headache | 16 | 11 | 19 | 19 | 19 | 19
  Malaise: number analyzed (Participants) | 73 | 71 | 73 | 71 | 72 | 68
  Malaise | 18 | 9 | 16 | 19 | 23 | 15
  Myalgia: number analyzed (Participants) | 73 | 71 | 73 | 71 | 72 | 68
  Myalgia | 32 | 29 | 35 | 36 | 39 | 28

3. Primary Outcome: Number of Participants With Solicited Injections Site or Systemic Reactions Following Vaccination at Day 0: Aged >=65 Years
Description: as for outcome 2
Time Frame: Within 7 days after vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Older Adults: SP0173 Formulation 4: Healthy participants aged >=65 years received a single dose of the SP0173 Tdap vaccine.
Arm/Group | Older Adults: SP0173 Formulation 1 | Older Adults: SP0173 Formulation 2 | Older Adults: SP0173 Formulation 3 | Older Adults: SP0173 Formulation 4 | Older Adults: Adacel® | Older Adults: Boostrix®
Number analyzed (Participants) | 77 | 73 | 78 | 72 | 76 | 78
Participants
  Injection site pain: number analyzed (Participants) | 77 | 73 | 78 | 72 | 75 | 78
  Injection site pain | 21 | 34 | 34 | 34 | 28 | 25
  Injection site erythema: number analyzed (Participants) | 77 | 73 | 78 | 72 | 75 | 78
  Injection site erythema | 0 | 1 | 2 | 2 | 3 | 1
  Injection site swelling: number analyzed (Participants) | 77 | 73 | 78 | 72 | 75 | 78
  Injection site swelling | 1 | 6 | 6 | 2 | 1 | 2
  Upper limb edema: number analyzed (Participants) | 75 | 70 | 75 | 71 | 72 | 74
  Upper limb edema | 38 | 43 | 36 | 38 | 32 | 40
  Extensive limb swelling | 0 | 0 | 0 | 0 | 0 | 0
  Fever: number analyzed (Participants) | 76 | 72 | 77 | 71 | 72 | 74
  Fever | 0 | 1 | 0 | 0 | 0 | 0
  Headache: number analyzed (Participants) | 77 | 73 | 78 | 72 | 74 | 77
  Headache | 6 | 10 | 20 | 12 | 11 | 14
  Malaise: number analyzed (Participants) | 77 | 73 | 77 | 72 | 74 | 77
  Malaise | 6 | 12 | 14 | 9 | 8 | 6
  Myalgia: number analyzed (Participants) | 77 | 73 | 77 | 72 | 74 | 77
  Myalgia | 12 | 21 | 30 | 23 | 23 | 17

ADVERSE EVENTS:
Time Frame: Non-serious AEs were collected from Day 0 to Day 7 (SRs) or Day 30 (unsolicited AEs) after vaccination. Serious AEs were collected from Day 0 up to Month 6 after vaccination.
Description: A SR was an AE that was prelisted (i.e. solicited) in the eCRF and considered to be related to vaccination (ADR). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. AEs were summarized in the safety analysis set.
Groups:
- Older Adults: SP0173 Formulation 1; Older Adults: SP0173 Formulation 2; Older Adults: SP0173 Formulation 3; Older Adults: SP0173 Formulation 4: Healthy participants aged >= 65 years received a single dose of the SP0173 Tdap vaccine.
- Older Adults: Adacel®: Healthy participants aged >= 65 years received Adacel®.
- Older Adults: Boostrix®: Healthy participants aged >= 65 years received Boostrix®.
Arm/Group | Adolescents: SP0173 Formulation 1 | Adolescents: SP0173 Formulation 2 | Adolescents: SP0173 Formulation 3 | Adolescents: SP0173 Formulation 4 | Adolescents: Adacel® | Adolescents: Boostrix® | Adults: SP0173 Formulation 1 | Adults: SP0173 Formulation 2 | Adults: SP0173 Formulation 3 | Adults: SP0173 Formulation 4 | Adults: Adacel® | Adults: Boostrix® | Older Adults: SP0173 Formulation 1 | Older Adults: SP0173 Formulation 2 | Older Adults: SP0173 Formulation 3 | Older Adults: SP0173 Formulation 4 | Older Adults: Adacel® | Older Adults: Boostrix®
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/71 | 0/77 | 0/77 | 0/75 | 0/75 | 0/76 | 0/73 | 0/76 | 0/76 | 0/76 | 1/72 | 0/77 | 0/73 | 0/78 | 0/72 | 0/76 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/71 | 0/77 | 1/77 | 0/75 | 0/75 | 1/76 | 1/73 | 1/76 | 1/76 | 0/76 | 2/72 | 0/77 | 3/73 | 4/78 | 1/72 | 2/76 | 2/78
Other Adverse Events (participants affected / at risk) | 71/79 | 64/71 | 67/77 | 68/77 | 71/75 | 66/75 | 52/76 | 53/73 | 67/76 | 54/76 | 62/76 | 50/72 | 53/77 | 60/73 | 58/78 | 53/72 | 49/76 | 56/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents: SP0173 Formulation 1 (N=79) | Adolescents: SP0173 Formulation 2 (N=71) | Adolescents: SP0173 Formulation 3 (N=77) | Adolescents: SP0173 Formulation 4 (N=77) | Adolescents: Adacel® (N=75) | Adolescents: Boostrix® (N=75) | Adults: SP0173 Formulation 1 (N=76) | Adults: SP0173 Formulation 2 (N=73) | Adults: SP0173 Formulation 3 (N=76) | Adults: SP0173 Formulation 4 (N=76) | Adults: Adacel® (N=76) | Adults: Boostrix® (N=72) | Older Adults: SP0173 Formulation 1 (N=77) | Older Adults: SP0173 Formulation 2 (N=73) | Older Adults: SP0173 Formulation 3 (N=78) | Older Adults: SP0173 Formulation 4 (N=72) | Older Adults: Adacel® (N=76) | Older Adults: Boostrix® (N=78)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device Dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug Withdrawal Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis Perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolic Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic Stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents: SP0173 Formulation 1 (N=79) | Adolescents: SP0173 Formulation 2 (N=71) | Adolescents: SP0173 Formulation 3 (N=77) | Adolescents: SP0173 Formulation 4 (N=77) | Adolescents: Adacel® (N=75) | Adolescents: Boostrix® (N=75) | Adults: SP0173 Formulation 1 (N=76) | Adults: SP0173 Formulation 2 (N=73) | Adults: SP0173 Formulation 3 (N=76) | Adults: SP0173 Formulation 4 (N=76) | Adults: Adacel® (N=76) | Adults: Boostrix® (N=72) | Older Adults: SP0173 Formulation 1 (N=77) | Older Adults: SP0173 Formulation 2 (N=73) | Older Adults: SP0173 Formulation 3 (N=78) | Older Adults: SP0173 Formulation 4 (N=72) | Older Adults: Adacel® (N=76) | Older Adults: Boostrix® (N=78)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change In Limb Circumference (General disorders) | 45 (45) | 41 (41) | 49 (49) | 46 (46) | 48 (48) | 33 (33) | 28 (28) | 37 (37) | 41 (41) | 37 (37) | 35 (35) | 31 (31) | 38 (38) | 43 (43) | 36 (36) | 38 (38) | 32 (32) | 40 (40)
Injection Site Erythema (General disorders) | 9 (9) | 4 (4) | 10 (10) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Injection Site Pain (General disorders) | 59 (59) | 51 (51) | 50 (50) | 49 (49) | 59 (59) | 48 (48) | 38 (38) | 34 (34) | 49 (49) | 42 (42) | 49 (49) | 35 (35) | 22 (22) | 34 (34) | 34 (34) | 34 (34) | 28 (28) | 25 (25)
Injection Site Swelling (General disorders) | 7 (7) | 4 (4) | 8 (8) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 6 (6) | 6 (6) | 2 (2) | 1 (1) | 2 (2)
Malaise (General disorders) | 14 (14) | 17 (17) | 14 (14) | 18 (18) | 12 (12) | 17 (17) | 18 (18) | 9 (9) | 16 (16) | 19 (19) | 23 (23) | 15 (15) | 6 (6) | 12 (12) | 14 (14) | 9 (9) | 8 (8) | 6 (6)
Pharyngitis (Infections and infestations) | 3 (3) | 7 (10) | 3 (3) | 5 (5) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 5 (5) | 4 (4) | 5 (7) | 5 (5) | 2 (2) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Pharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 42 (42) | 35 (35) | 38 (38) | 42 (42) | 52 (52) | 38 (38) | 32 (32) | 29 (29) | 35 (35) | 36 (36) | 39 (39) | 28 (28) | 12 (12) | 21 (21) | 31 (31) | 23 (23) | 23 (23) | 18 (18)
Headache (Nervous system disorders) | 23 (25) | 15 (15) | 19 (21) | 25 (26) | 22 (22) | 29 (30) | 16 (16) | 11 (11) | 19 (19) | 19 (19) | 19 (19) | 19 (21) | 6 (6) | 10 (10) | 20 (20) | 12 (12) | 11 (11) | 14 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 4 (4) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 2 (2) | 2 (2) | 4 (5) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT02587520/Prot_001.pdf
  • Statistical Analysis Plan (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT02587520/SAP_000.pdf